CLINICAL TRIAL: NCT04912986
Title: Construction and Application of Early Lung Rehabilitation Training Programs for Adult Patients After Double Lung Transplantation
Brief Title: Construction and Application of Early Lung Rehabilitation Training Programs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0232
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Transplantation
Keywords: pulmonary transplantation; pulmonory rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment (Placebo Comparator): Review the collection of patient-related clinical data, collation of clinical data and outcome indicators
  Interventions: Behavioral: Routine treatment
- Experimental group (Experimental): The intervention was implemented in accordance with the Early Lung Rehabilitation Training Programme for Adult Double Lung Transplant Patients
  Interventions: Behavioral: Early Lung Rehabilitation Training

INTERVENTIONS:
Behavioral: Early Lung Rehabilitation Training — It is implemented in accordance with the Early Lung Rehabilitation Training Program for Adult Double Lung Transplant Patients. Establish multidisciplinary collaboration teams, including competent doctors, nurses, rehabilitation physicians, and psychologists.
  Arms: Experimental group
Behavioral: Routine treatment — Provide rehabilitation training as usual, without standard program
  Arms: routine treatment

SUMMARY:
This study is intended to construct early lung rehabilitation training programs for adult patients after double lung transplantation, including safety assessment, exercise training, respiratory function training, psychological support and health education, with a view to helping double lung transplant patients achieve lung rehabilitation at an early date, improve patients' motor endurance and respiratory function, and improve the quality of near- and long-term survival.

DETAILED DESCRIPTION:
The first stage constructs the lung rehabilitation program, and the second stage implements the non-contemporaneous study control trial.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* consent to early lung rehabilitation
* informed consent to this study.

Exclusion Criteria:

* Unstable condition, not allowed to receive pulmonary rehabilitation treatment
* A person with a mental disorder who cannot cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation time | 1 year
  The time for mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jiangshuyuan Liang, Master, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No